CLINICAL TRIAL: NCT00712881
Title: Prospective, Open-Label, Randomized Study of Combination Therapy of MYOCET® Plus Cyclophosphamide and Trastuzumab Versus Free Doxorubicin Plus Cyclophosphamide Alone, Each Followed by Docetaxel and Trastuzumab, in Neoadjuvant Setting in Treatment-Naive Patients With HER2-Positive Breast Cancer
Brief Title: Combination Therapy With MYOCET® (Doxorubicin HCL Liposome for Injection) in Participants With HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C19562/2037; 2008-000709-12 (EudraCT Number)
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Trastuzumab; Anthracyclines; Docetaxel

ARMS (2):
- Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) (Experimental): Participants will receive MCH (liposomal doxorubicin hydrochloride [60 milligrams {mg}/square meter {m^2}], cyclophosphamide (600 mg/m^2), and trastuzumab (8 or 6 mg/kilogram {kg}), administered as intravenous (IV) infusion on Day 1 of each of 4 consecutive 21-day cycles. For the first cycle, the loading dose of trastuzumab will be 8 mg/kg; 6 mg/kg will be used for the remaining cycles. After 4 cycles of MCH, the treatment will be changed to 4 consecutive 21-day cycles of TH (docetaxel [100 mg/m^2] and trastuzumab [6 mg/kg]).
  Interventions: Drug: Liposomal doxorubicin hydrochloride; Drug: Cyclophosphamide; Drug: Trastuzumab; Drug: Docetaxel
- Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH) (Active Comparator): Participants will receive AC (free doxorubicin hydrochloride [60 mg/m^2] and cyclophosphamide [600 mg/m^2]), administered as IV infusion on Day 1 of each of 4 consecutive 21-day cycles. After 4 cycles of AC, the treatment will be changed to 4 consecutive 21-day cycles of TH (docetaxel [100 mg/m^2] and trastuzumab [8 or 6 mg/kg]). For the first cycle, the loading dose of trastuzumab will be 8 mg/kg; 6 mg/kg will be used for the remaining cycles.
  Interventions: Drug: Cyclophosphamide; Drug: Trastuzumab; Drug: Free doxorubicin hydrochloride; Drug: Docetaxel

INTERVENTIONS:
Drug: Liposomal doxorubicin hydrochloride — Liposomal doxorubicin hydrochloride will be administered per dose and schedule specified in the arm description.
  Other Names: Myocet®
  Arms: Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH)
Drug: Cyclophosphamide — Cyclophosphamide will be administered per dose and schedule specified in the arm description.
Drug: Trastuzumab — Trastuzumab will be administered per dose and schedule specified in the arm description.
Drug: Free doxorubicin hydrochloride — Free doxorubicin hydrochloride will be administered per dose and schedule specified in the arm description.
  Other Names: Anthracycline
  Arms: Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH)
Drug: Docetaxel — Docetaxel will be administered per dose and schedule specified in the arm description.

SUMMARY:
To evaluate the efficacy and safety of treatment with MYOCET® (doxorubicin hydrochloride) in combination with cyclophosphamide and trastuzumab, 4 cycles, followed by docetaxel plus trastuzumab, 4 cycles, in women with stage II or III breast cancer whose tumour overexpresses the human epidermal growth factor receptor 2 (HER2) gene.

ELIGIBILITY:
Main Inclusion Criteria:

* Treatment-naive participants with stage II or III invasive breast cancer (proven histologically/cytologically) and with tests showing an overexpressing of HER2.
* Participants have at least 1 bidimensionally measurable lesion according to the World Health Organization (WHO) criteria.
* The participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The participant has an LVEF of at least 55% as assessed by multigated acquisition (MUGA) scan (preferred) or echocardiography.
* The participant has hematology and serum chemistry laboratory test results within specific protocol-defined ranges.
* Women of childbearing potential must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the treatment period and for 6 months after the last administration of study drug.

Main Exclusion Criteria:

The participant:

* Has received previous cancer therapy for breast cancer.
* Has any history of CHF, angina pectoris, or myocardial infarction.
* Has uncontrolled hypertension.
* Has infection, peptic ulcer, or unstable diabetes mellitus.
* Has been treated with live virus vaccines within 8 weeks before the first administration of study drug.
* Has impaired hepatic or renal function.
* Is a pregnant or lactating woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
* Has used an investigational drug within one month before the screening visit.
* Has a known hypersensitivity to any of the study drugs or to their active ingredients.
* Has an inflammatory breast cancer.
* Has had any other malignancies within five years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer).

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-10-13 (Actual); Primary Completion 2015-09-17 (Actual); Study Completion 2015-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (22):
- Austria (2):
  - Teva Investigational Site 16, Kufstein
  - Teva Investigational Site 15, Vienna
- Belgium (2):
  - Teva Investigational Site 9, Brussels
  - Teva Investigational Site 29, Yvoir
- France (4):
  - Teva Investigational Site 4, Clichy
  - Teva Investigational Site 5, Nancy
  - Teva Investigational Site 33, Reims
  - Teva Investigational Site 8, Vandœuvre-lès-Nancy
- Germany (7):
  - Teva Investigational Site 30, Aachen
  - Teva Investigational Site 11, Düsseldorf
  - Teva Investigational Site 25, Düsseldorf
  - Teva Investigational Site 32, Essen
  - Teva Investigational Site 34, Loerrach
  - Teva Investigational Site 14, München
  - Teva Investigational Site 27, München
- Italy (3):
  - Teva Investigational Site 20, Napoli
  - Teva Investigational Site 23, Roma
  - Teva Investigational Site 21, Verona
- Spain (4):
  - Teva Investigational Site 26, Barcelona
  - Teva Investigational Site 3, Barcelona
  - Teva Investigational Site 1, Lleida
  - Teva Investigational Site 2, Zaragoza

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned in 1:1 ratio to investigational group (Doxorubicin [MYOCET] + Cyclophosphamide + Trastuzumab [MCH] and Docetaxel + Trastuzumab [TH]) and comparison group (Doxorubicin [Anthracycline] + Cyclophosphamide [AC] and Docetaxel + Trastuzumab [TH]).
Groups:
- Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH): Participants received MCH (liposomal doxorubicin hydrochloride [60 milligrams {mg}/square meter {m^2}], cyclophosphamide (600 mg/m^2), and trastuzumab (8 or 6 mg/kilogram {kg}), administered as intravenous (IV) infusion on Day 1 of each of 4 consecutive 21-day cycles. For the first cycle, the loading dose of trastuzumab was 8 mg/kg; 6 mg/kg was used for the remaining cycles. After 4 cycles of MCH, the treatment changed to 4 consecutive 21-day cycles of TH (docetaxel [100 mg/m^2] and trastuzumab [6 mg/kg]).
- Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH): Participants received AC (free doxorubicin hydrochloride [60 mg/m^2] and cyclophosphamide [600 mg/m^2]), administered as IV infusion on Day 1 of each of 4 consecutive 21-day cycles. After 4 cycles of AC, the treatment changed to 4 consecutive 21-day cycles of TH (docetaxel [100 mg/m^2] and trastuzumab [8 or 6 mg/kg]). For the first cycle, the loading dose of trastuzumab was 8 mg/kg; 6 mg/kg was used for the remaining cycles.
Period: Overall Study
Arm/Group | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH)
Started | 63 | 63
Received at Least 1 Dose of Study Drug | 62 | 63
Completed 8 Cycles of Treatment | 55 | 56
Completed | 53 | 56
Not Completed | 10 | 7
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Disease Progression | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Non-Compliance To Study Procedures | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Randomized but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: The set of enrolled participants included all participants who were randomized to a treatment group, regardless of whether or not a participant received any study drug.
Groups:
- Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH): Participants received MCH (liposomal doxorubicin hydrochloride [60 mg/m^2], cyclophosphamide (600 mg/m^2), and trastuzumab (8 or 6 mg/kg), administered as IV infusion on Day 1 of each of 4 consecutive 21-day cycles. For the first cycle, the loading dose of trastuzumab was 8 mg/kg; 6 mg/kg was used for the remaining cycles. After 4 cycles of MCH, the treatment changed to 4 consecutive 21-day cycles of TH (docetaxel [100 mg/m^2] and trastuzumab [6 mg/kg]).
- Total: Total of all reporting groups
Arm/Group | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH) | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (11.6) | 51.1 (11.3) | 49.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 63 | 126
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 61 | 59 | 120
  Black | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Other | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Exhibiting a Pathological Complete Response (pCR) in Breast
Description: The pCR of breast was based upon histologic examination, as confirmed by a central panel of experts, of resected tissue .
Time Frame: At the end of Cycle 8 (each cycle length = 21 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH)
Number analyzed (Participants) | 63 | 63
percentage of participants | 41.3 | 54.0
Statistical Analysis 1: Comparison: Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) vs Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH); Test type: Other; p = 0.154, 2-sided, binomial proportions — Threshold for significance at 0.05 level

2. Secondary Outcome: Percentage of Participants Who Achieved an Objective Response (Complete Response [CR] or Partial Response [PR]), as Defined by World Health Organization (WHO) Guidelines
Description: CR: Disappearance of the lesions and no new lesions. In case of bone metastasis a CR is represented by the normalization of radiography or the complete sclerotic healing of lytic area.
  PR: In the case of bidimensionally measurable lesions/tumors, a decrease by at least 50% of the sum of the products of the largest perpendicular diameters of each individual lesion/tumor. In the case of unidimensionally measurable lesions a decrease by at least 50% in the largest linear tumour measurement. In the case of non-measurable but evaluable lesions an appreciable change of lesions referable to disease improvement. For bone lesions partial decrease in size or recalcification of lytic areas. No lesion should have progressed and no new lesion should appear.
Time Frame: At the end of Cycle 8 (each cycle length = 21 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH)
Number analyzed (Participants) | 63 | 63
percentage of participants | 77.8 | 84.1

3. Secondary Outcome: Percentage of Participants With Class III or IV New York Health Association (NYHA) Congestive Heart Failure (CHF)
Description: Occurrence of Class III or IV (NYHA) CHF has been reported. Class III: Participants with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain. Class IV: Participants with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: Baseline up to the end of Cycle 8 (each cycle length = 21 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH)
Number analyzed (Participants) | 63 | 63
percentage of participants | 0 | 0

4. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF)
Description: The LVEF is a fraction of blood (in percent) pumped out of the left ventricle of the heart (the main pumping chamber). LVEF was measured using multigated acquisition (MUGA) or echocardiography.
Time Frame: Baseline, up to 5 years
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug. Here, 'Number analyzed' = participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: percentage of blood pumped out
Arm/Group | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH)
Number analyzed (Participants) | 62 | 63
percentage of blood pumped out
  Change at Cycle 4: number analyzed (Participants) | 54 | 56
  Change at Cycle 4 | -1.5 (6.5) | -1.0 (5.3)
  Change at Pre-surgery Visit: number analyzed (Participants) | 45 | 47
  Change at Pre-surgery Visit | -0.8 (7.1) | -3.4 (6.4)
  Change at Post-surgery Visit: number analyzed (Participants) | 29 | 29
  Change at Post-surgery Visit | -1.6 (7.3) | -3.6 (5.7)
  Change at Month 12: number analyzed (Participants) | 50 | 54
  Change at Month 12 | -0.9 (7.0) | -4.4 (8.0)
  Change at Month 24: number analyzed (Participants) | 41 | 41
  Change at Month 24 | 0.6 (8.0) | -4.7 (7.9)
  Change at Month 36: number analyzed (Participants) | 31 | 28
  Change at Month 36 | 2.1 (5.6) | -3.8 (7.4)
  Change at Month 48: number analyzed (Participants) | 31 | 27
  Change at Month 48 | -1.3 (8.3) | -2.5 (9.0)
  Change at Month 60: number analyzed (Participants) | 23 | 25
  Change at Month 60 | -1.0 (7.7) | -1.4 (11.0)

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. The TEAE was an AE that began or worsened after treatment with study drug. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline up to the end of Cycle 8 (cycle length = 21 days)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH)
Number analyzed (Participants) | 62 | 63
Participants | 62 | 63

6. Secondary Outcome: Percentage of Participants With Progression or Death
Description: Progression was defined as a 25% or more increase in the size of the lesion or appearance of new lesion. If the participant did not develop an event (disease progression or death), the participant was censored at the last known tumor assessment date (or last follow-up visit without progression documented).
Time Frame: Up to 5 Years after randomization
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH)
Number analyzed (Participants) | 63 | 63
percentage of participants
  Participants with progression or death | 11.1 | 12.7
  Participants censored | 88.9 | 87.3

7. Secondary Outcome: Percentage of Participants Achieving a Pathological Complete Response (pCR) in Breast and Node
Description: The pCR of breast and node was based upon histologic examination, as confirmed by a central panel of experts, of breast tissue resected.
Time Frame: At the end of Cycle 8 (each cycle length = 21 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH)
Number analyzed (Participants) | 63 | 63
percentage of participants | 38.1 | 47.6

8. Secondary Outcome: Number of Participants Undergoing Breast Conservative Surgery
Time Frame: At the end of Cycle 8 (each cycle length = 21 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH)
Number analyzed (Participants) | 63 | 63
Participants
  Missing data | 7 | 5
  Had breast conservative surgery | 33 | 31
  Did not have breast conservative surgery | 23 | 27

9. Secondary Outcome: Severity of Adverse Events as Characterized by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Description: AEs were recorded and graded per the NCI CTCAE scale. The NCI CTCAE is a toxicity scale used to grade the severity of adverse events experienced with cancer treatment. Grade 1= Mild; Grade 2= Moderate; Grade 3= Severe; Grade 4= Life-threatening or disabling; Grade 5= Death related to AE. For summaries for the toxicity grade, participants were counted once at the greatest NCI CTCAE grade.
Time Frame: Up to Week 24
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH)
Number analyzed (Participants) | 62 | 63
Participants
  Grade 1 | 2 | 1
  Grade 2 | 9 | 12
  Grade 3 | 19 | 18
  Grade 4 | 32 | 32
  Grade 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years after randomization
Description: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH)
All-Cause Mortality (participants affected / at risk) | 0/62 | 4/63
Serious Adverse Events (participants affected / at risk) | 18/62 | 21/63
Other Adverse Events (participants affected / at risk) | 62/62 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) (N=62) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH) (N=63)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9) | 7 (7)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Whiplash injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 1 (2) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin (MYOCET) + Cyclophosphamide + Trastuzumab (MCH) and Docetaxel + Trastuzumab (TH) (N=62) | Doxorubicin (Anthracycline) + Cyclophosphamide (AC) and Docetaxel + Trastuzumab (TH) (N=63)
Anaemia (Blood and lymphatic system disorders) | 13 (27) | 21 (60)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 24 (77) | 34 (111)
Lymphopenia (Blood and lymphatic system disorders) | 3 (15) | 6 (17)
Neutropenia (Blood and lymphatic system disorders) | 41 (145) | 46 (143)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 5 (8)
Vertigo (Ear and labyrinth disorders) | 5 (8) | 5 (6)
Conjunctivitis (Eye disorders) | 11 (12) | 10 (13)
Lacrimation increased (Eye disorders) | 6 (7) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 5 (8) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 12 (19) | 12 (16)
Constipation (Gastrointestinal disorders) | 19 (35) | 16 (28)
Diarrhoea (Gastrointestinal disorders) | 27 (57) | 25 (44)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 8 (9) | 9 (10)
Nausea (Gastrointestinal disorders) | 44 (95) | 39 (95)
Stomatitis (Gastrointestinal disorders) | 21 (47) | 21 (45)
Vomiting (Gastrointestinal disorders) | 17 (29) | 21 (38)
Asthenia (General disorders) | 28 (115) | 36 (116)
Fatigue (General disorders) | 19 (51) | 15 (54)
Infusion related reaction (General disorders) | 3 (5) | 4 (4)
Mucosal inflammation (General disorders) | 32 (62) | 25 (55)
Oedema (General disorders) | 10 (13) | 7 (9)
Oedema peripheral (General disorders) | 9 (10) | 11 (15)
Pain (General disorders) | 1 (2) | 4 (5)
Pyrexia (General disorders) | 17 (21) | 11 (21)
Bronchitis (Infections and infestations) | 3 (4) | 4 (7)
Nasopharyngitis (Infections and infestations) | 4 (6) | 16 (21)
Respiratory tract infection (Infections and infestations) | 4 (4) | 4 (5)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 4 (7) | 0 (0)
Alanine aminotransferase increased (Investigations) | 10 (17) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 6 (8) | 5 (6)
Blood lactate dehydrogenase increased (Investigations) | 4 (4) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 10 (18) | 4 (4)
Weight increased (Investigations) | 0 (0) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 12 (16) | 12 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (16) | 10 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 18 (28) | 15 (33)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 (35) | 13 (36)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (26) | 17 (23)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (2)
Disturbance in attention (Nervous system disorders) | 4 (5) | 3 (4)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3)
Dysgeusia (Nervous system disorders) | 14 (24) | 13 (15)
Headache (Nervous system disorders) | 13 (20) | 15 (20)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 7 (9)
Neurotoxicity (Nervous system disorders) | 1 (1) | 4 (6)
Paraesthesia (Nervous system disorders) | 9 (14) | 15 (31)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (14) | 2 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 5 (5)
Depression (Psychiatric disorders) | 4 (4) | 3 (4)
Insomnia (Psychiatric disorders) | 7 (10) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 8 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 6 (6)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 37 (55) | 41 (52)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (17) | 7 (8)
Erythema (Skin and subcutaneous tissue disorders) | 6 (8) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 13 (19) | 11 (13)
Nail toxicity (Skin and subcutaneous tissue disorders) | 8 (11) | 6 (7)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 (13) | 7 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 11 (16) | 8 (14)
Skin toxicity (Skin and subcutaneous tissue disorders) | 10 (11) | 4 (8)
Hot flush (Vascular disorders) | 10 (12) | 12 (20)
Hypertension (Vascular disorders) | 3 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.